CLINICAL TRIAL: NCT06988033
Title: Effects of Different Vibration Applications on Bone Turnover Markers and Functionality After Total Knee Arthroplasty in Women With Osteopenia: A Randomized Controlled Trial
Brief Title: Vibration Applications After Total Knee Arthroplasty in Osteopenic Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstinyeUni-EALOGLUCIFTCI-001
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Osteopenia; Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Osteopenia; Vibration; Women; Bone Turnover Markers
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel arms: Whole Body Vibration (WBV), WBV with exercise, or Control (standard rehabilitation). Each arm will receive a distinct intervention protocol concurrently over the same study period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole Body Vibration (Experimental): Participants in this group will receive whole body vibration (WBV) in addition to the standard postoperative rehabilitation program. WBV will be applied 3 times per week. In the first week, 1 set of 5-minute static standing WBV will be administered at a low frequency (8 Hz) and amplitude (2 mm). In subsequent weeks, progression will be applied based on participant tolerance. The frequency will increase gradually up to 30-40 Hz, and the amplitude up to 5 mm, with a total WBV duration of up to 15 minutes per session. Participants will stand upright with equal weight distribution on both feet during vibration. No concurrent exercise will be performed during WBV.
  Interventions: Behavioral: Whole Body Vibration Therapy
- Whole Body Vibration with Exercise (WBV-E) (Experimental): In this group, participants will receive whole body vibration (WBV) simultaneously with lower extremity exercises performed on a vibrating platform. After exercise training is demonstrated on a stable surface, participants will perform the exercises on the platform. WBV will be initiated with low amplitude (2 mm) for the first two weeks and increased to 5 mm by the third week depending on pain tolerance. Frequency will be maintained between 30-40 Hz. Exercises will include lunge steps, shallow squats, dynamic squats, toe raises, and ball squeezes between the knees (2-3 kg medicine ball). Vibration duration will progress from 2 minutes (3 exercises × 30 sec) to a maximum of 18 minutes (6 exercises × 60 sec × 3 sets). One-minute rest will be provided between sets and repetitions. Total session duration will vary between 45 and 70 minutes.
  Interventions: Behavioral: Whole Body Vibration with Exercise
- Control (Active Comparator): Participants in this group will receive only the standard postoperative rehabilitation program and an individualized home exercise plan. The conventional rehabilitation protocol includes exercises with rest periods of 1 minute between sets and repetitions. The average initial session duration will be approximately 45 minutes, progressing to 60-70 minutes in later sessions. No vibration intervention will be administered.
  Interventions: Behavioral: Conventional Physiotherapy

INTERVENTIONS:
Behavioral: Whole Body Vibration Therapy — Participants receive whole-body vibration therapy in a static upright position on a vibration platform (Power Plate My5). The intervention is applied 3 times per week for 8 weeks, progressively increasing frequency from 8 Hz to 40 Hz and amplitude from 2 mm to 5 mm. Each session lasts up to 15 minutes. No exercise is performed during the vibration.
  Arms: Whole Body Vibration
Behavioral: Whole Body Vibration with Exercise — Participants perform lower extremity strengthening exercises on a vibration platform simultaneously with whole-body vibration. The protocol includes lunges, squats, heel raises, and ball squeezes. Vibration frequency ranges from 30 to 40 Hz and amplitude from 2 to 5 mm. Sessions are performed 3 times per week for 8 weeks, with duration progressing from 2 to 18 minutes depending on tolerance.
  Arms: Whole Body Vibration with Exercise (WBV-E)
Behavioral: Conventional Physiotherapy — Participants receive standard post-total knee arthroplasty physiotherapy 3 times per week for 12 weeks, lasting 40 to 70 minutes per session. In addition, a home-based exercise program is performed 3 times daily. The program includes range of motion, strengthening, and balance exercises. No vibration therapy is applied in this group.
  Arms: Control

SUMMARY:
Osteoarthritis (OA) is a chronic degenerative disease characterized by the destruction of articular cartilage, leading to functional impairment of surrounding bone and soft tissues. It is a major global public health problem, with the knee joint being the most commonly affected site. Treatment modalities include exercise, diet, oral non-steroidal anti-inflammatory drugs (NSAIDs), intra-articular injections, and total knee arthroplasty (TKA). TKA is indicated in cases of severe pain, functional loss, deformity, and limited range of motion when conservative methods are no longer effective. However, some patients may continue to experience deformity and functional deficits after surgery. Postoperative quadriceps weakness and decreased functional capacity can negatively affect patient prognosis.

Following TKA, bone mineral density (BMD) tends to decrease during the first three months. The reduction in BMD and the increase in bone resorption may elevate the risk of implant loosening or periprosthetic fracture. Bone turnover markers (BTMs), which are enzymes or degradation products released into circulation by bone cells, reflect bone remodeling processes and can help identify increased fracture risk.

A significant proportion of TKA candidates are osteopenic. Since osteopenic individuals make up a larger segment of the population, most fragility fractures actually occur in individuals with osteopenia rather than osteoporosis. Therefore, BMD levels and the presence of osteopenia or osteoporosis should be taken into account in patients undergoing TKA.

To preserve both bone quality and muscle mass, early rehabilitation and progressive weight-bearing on the operated limb are considered essential. These strategies may improve both BMD and BTMs. Whole-body vibration (WBV) therapy has been suggested as an effective and safe method to increase mechanical loading on the bones. WBV can be applied in a static standing position on a vibration platform or combined with simultaneous exercise.

Given the limited availability of targeted strategies to improve bone remodeling and BTMs after TKA, and the lack of clarity regarding the optimal WBV protocol, this study aims to investigate the effects of different vibration applications on bone turnover markers, functionality, muscle strength, pain intensity, pressure pain threshold, range of motion, proprioception, edema, and muscle biomechanical properties in osteopenic women following TKA.

Participants will be randomly assigned to one of three groups: WBV only, WBV combined with exercise (WBV-E), or control. All groups will receive traditional rehabilitation three times per week for four weeks after surgery. WBV interventions will begin at the end of the fourth postoperative week, once patients are deemed ready. While WBV groups will receive additional vibration therapy, the control group will continue traditional rehabilitation alone.

Outcomes will be evaluated using bone turnover markers, the Timed Up and Go (TUG) test, the 30-Second Chair Stand Test, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), measurements of muscle biomechanical properties and strength, pain intensity and pressure pain threshold, joint range of motion, proprioception, and edema.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo unilateral, primary, cemented total knee arthroplasty (TKA) using a posterior cruciate ligament-sacrificing technique and medial parapatellar approach due to knee osteoarthritis
* Ability to speak and understand Turkish
* Ability to comprehend both verbal and written information
* A T-score between -2.5 and -1 (i.e., -2.5 < T-score < -1) measured by DXA in the lumbar spine, total hip, or femoral neck within the past year

Exclusion Criteria:

* Scheduled for revision TKA
* American Society of Anesthesiologists (ASA) physical status classification score higher than 3
* History of major surgery on the limb to be operated
* Presence of comorbid diseases such as rheumatoid arthritis or cancer
* Presence of a neurological condition causing functional impairment
* Diagnosed psychiatric disorder
* Dementia
* Disorders affecting the vestibular system
* Having undergone anesthesia for any reason within the last month
* Regular use of hypnotic or anxiolytic medications
* Hearing or vision impairment not correctable by hearing aids or glasses
* Presence of endocrine system disorders
* Secondary osteoporosis or history of osteoporotic fracture
* Metabolic bone diseases or chronic illnesses potentially affecting bone metabolism
* Use of medications known to affect bone metabolism (e.g., menopausal hormone therapy, bisphosphonates, raloxifene, calcitonin, growth hormone, parathyroid hormones, corticosteroids) within 6 months prior to the start of the study

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) Test Score | Baseline (Week 4 post-op) and 12th week (Post-intervention)
  This test evaluates functional mobility and performance-based activity limitation. Participants are instructed to stand up from a standardized chair (height: 44 cm; depth: 26 cm), walk 3 meters at a normal pace, turn around, return, and sit down. The time taken to complete the task is recorded. The TUG test is a valid and reliable indicator of physical function in individuals with knee osteoarthritis.
Bone Turnover Marker (Serum Procollagen Type I N-terminal Propeptide (PINP) Level) | Pre-surgery, Week 4, Week 12
  Serum PINP levels will be measured using enzyme-linked immunosorbent assay (ELISA) to evaluate bone formation activity. Results will be expressed in nanograms per milliliter (ng/mL). Blood samples will be collected at three time points: pre-surgery, week 4 post-surgery, and week 12 post-surgery
Bone Turnover Marker (Serum Osteocalcin (OCN) Level) | Pre-surgery, Week 4, Week 12
  Serum concentration of Osteocalcin (OCN )will be measured using enzyme-linked immunosorbent assay (ELISA) to evaluate bone turnover. Units will be expressed in nanograms per milliliter (ng/mL). Blood samples will be collected at 3 time points: pre-surgery, week 4, and week 12 post-surgery.
Bone Turnover Marker (Serum C-terminal Telopeptide of Type I Collagen (CTX) Level) | Pre-surgery, Week 4, Week 12
  C-terminal Telopeptide of Type I Collagen (CTX) concentrations will be analyzed using enzyme-linked immunosorbent assay (ELISA) to evaluate bone resorption. Results will be expressed in nanograms per milliliter (ng/mL). Serum will be collected at three time points: before surgery, and at 4 and 12 weeks after surgery.
Bone Turnover Marker (Serum N-terminal Telopeptide of Type I Collagen (NTX) Level) | Pre-surgery, Week 4, Week 12
  N-terminal Telopeptide of Type I Collagen (NTX) will be measured with enzyme-linked immunosorbent assay (ELISA) kits to assess bone resorption activity. Results will be expressed in nanomoles of bone collagen equivalents per liter (nmol BCE/L), according to kit instructions. Samples will be drawn at three time points: pre-surgery, week 4, and week 12 post-surgery.
30-Second Chair Stand Test | Week 4 and Week 12
  Participants are asked to cross their arms over their chest and stand up from a 44 cm standard chair as many times as possible within 30 seconds. The number of correct repetitions is recorded to assess lower limb functional strength and endurance.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Week 4 and Week 12
  The WOMAC index evaluates pain, stiffness, and physical function through 24 items scored from 0 to 4. Higher scores indicate greater impairment.
Muscle Strength (Isometric) | Week 4 and Week 12
  Maximum isometric knee extension (quadriceps) strength will be assessed using a Lafayette digital dynamometer with standardized seated positioning (hip 90°, knee 60° flexion). The average of three trials will be recorded in Newton.
Pain Pressure Threshold (PPT) | Week 4 and Week 12
  Pressure pain threshold will be assessed using a 10-anatomical point digital pressure algometer (J-TECH-USA Commander) that has shown excellent relative and absolute reliability in knee osteoarthritis. Measurements will be recorded in kilogram-force (kg). The average value of the 10 anatomical points will be used for analysis.

SECONDARY OUTCOMES:
Pain Intensity (Visual Analog Scale) | Week 4 and Week 12
  Pain severity during rest, walking, and night will be measured using a 100-mm Visual Analog Scale (VAS). Higher scores represent more severe pain.
Knee Range of Motion (ROM) | Week 4 and Week 12
  Active and passive flexion and extension ROM of the knee will be measured using a Baseline goniometer. Values will be recorded in degrees.
Proprioception (Joint Position Sense) | Week 4 and Week 12
  Active joint position reproduction test at 30° and 60° knee flexion will be performed. The angular error from the target position will be measured using a goniometer. The mean of three trials will be calculated.
Knee Edema Volume | Week 4 and Week 12
  Edema volume will be calculated using circumferential measurements taken every 5 cm between 10 cm proximal and distal to the medial femoral condyle. Volume will be estimated using the Frustum formula.
Biomechanical Muscle Properties (Muscle Tone of Quadriceps) | Week 4 and Week 12
  Muscle tone (resting tension) of the quadriceps (vastus lateralis, vastus medialis, rectus femoris) will be measured using the MyotonPRO device. Measurements will be recorded in Hertz (Hz). Measurements will be made three times for each part of the muscle and the average value will be taken. Separate values will be recorded for vastus lateralis, vastus medialis, rectus femoris.
Biomechanical Muscle Properties (Muscle Stiffness of Quadriceps) | Week 4 and Week 12
  Muscle stiffness of the quadriceps (vastus lateralis, vastus medialis, rectus femoris) will be measured using the MyotonPRO device. Results will be reported in Newtons per meter (N/m). Measurements will be made three times for each part of the muscle and the average value will be taken. Separate values will be recorded for vastus lateralis, vastus medialis, rectus femoris.
Biomechanical Muscle Properties (Muscle Elasticity of Quadriceps) | Week 4 and Week 12
  Muscle elasticity will be characterized by the logarithmic decrement (D) measured using the MyotonPRO device. This is a unitless (relative) value representing the ability of the muscle to restore its shape after deformation. Measurements will be made three times for each part of the muscle and the average value will be taken. Separate values will be recorded for vastus lateralis, vastus medialis, rectus femoris.
Biomechanical Muscle Properties (Muscle Relaxation Time of Quadriceps) | Week 4 and Week 12
  Mechanical stress relaxation time (R) will be measured using the MyotonPRO to assess the time the muscle takes to return to rest following deformation. Results will be reported in milliseconds (ms). Measurements will be made three times for each part of the muscle and the average value will be taken. Separate values will be recorded for vastus lateralis, vastus medialis, rectus femoris.
Biomechanical Muscle Properties (Muscle Creep of Quadriceps) | Week 4 and Week 12
  Muscle creep will be assessed as the ratio of relaxation and deformation time (Creep (C)) using the MyotonPRO device. This parameter is a relative unit and indicates viscoelastic behavior of the muscle. Measurements will be made three times for each part of the muscle and the average value will be taken. Separate values will be recorded for vastus lateralis, vastus medialis, rectus femoris.

OTHER OUTCOMES:
Perceived Exertion Level (Borg-RPE15 Scale) | At each exercise session from Week 1 to Week 12
  Perceived exertion will be assessed to monitor exercise progression and evaluate effort intensity using the Borg Rating of Perceived Exertion Scale (Borg-RPE15). This scale is designed to measure the subjective level of exertion experienced by participants following strength training. The Borg-RPE15 ranges from 6 to 20, where a score of 6 indicates rest, 7-9 indicates light effort, 11-13 moderate effort, and 15 or above represents high-intensity exertion.

CONTACTS AND LOCATIONS:
Overall Officials: GÜL DENİZ YILMAZ YELVAR, ASSOCIATE PROFESSOR, Study Chair — Istinye University
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified, summary-level outcome data, including group-level means, standard deviations, effect sizes, and p-values derived from statistical analyses. These data will be provided to support transparency and allow for interpretation of the study findings.
Supporting Information: Study Protocol, SAP
Time Frame: Summary-level data and supporting documents (e.g., study protocol and statistical analysis plan) will be available within 12 months following the final publication of study results and will remain accessible for at least 5 years via institutional repository or upon reasonable request.
Access Criteria: The study's outcome results, including group-level means, standard deviations, p-values, and effect sizes, as well as supporting materials such as the study protocol and statistical analysis plan, will be made available to qualified academic researchers upon reasonable request. Data will be provided for ethically approved, non-commercial research purposes. Interested investigators should contact the principal investigator through the affiliated institution and submit a written request describing the intended use and data handling procedures. Each request will be reviewed individually in accordance with institutional data-sharing guidelines.

REFERENCES:
- [Background] He Z, Zheng J, Liu S, Guan Z, Zhou Q, Jin X, Guan Z. The effect of whole-body vibration in osteopenic patients after total knee arthroplasty: a randomized controlled trial. Aging Clin Exp Res. 2022 Jun;34(6):1381-1390. doi: 10.1007/s40520-021-02043-2. Epub 2022 Jan 14. PMID 35028919
- [Background] Gazdzik TS, Gajda T, Kaleta M. Bone mineral density changes after total knee arthroplasty: one-year follow-up. J Clin Densitom. 2008 Jul-Sep;11(3):345-50. doi: 10.1016/j.jocd.2008.04.007. Epub 2008 Jul 10. PMID 18619880
- [Background] Cardinale M, Bosco C. The use of vibration as an exercise intervention. Exerc Sport Sci Rev. 2003 Jan;31(1):3-7. doi: 10.1097/00003677-200301000-00002. PMID 12562163
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Klug A, Gramlich Y, Rudert M, Drees P, Hoffmann R, Weissenberger M, Kutzner KP. The projected volume of primary and revision total knee arthroplasty will place an immense burden on future health care systems over the next 30 years. Knee Surg Sports Traumatol Arthrosc. 2021 Oct;29(10):3287-3298. doi: 10.1007/s00167-020-06154-7. Epub 2020 Jul 15. PMID 32671435
- [Background] Sowers M. Epidemiology of risk factors for osteoarthritis: systemic factors. Curr Opin Rheumatol. 2001 Sep;13(5):447-51. doi: 10.1097/00002281-200109000-00018. PMID 11604603